CLINICAL TRIAL: NCT04331080
Title: A Phase 2b/3 Randomized, Prospective, Double Blind, Within-Subject Vehicle Controlled, Multi-Center Study to Determine the Efficacy and Safety of Granexin® Gel in Reducing Scar Formation in Surgical Wounds Following Bilateral Anchor Incision Breast Surgery
Brief Title: A Study of Granexin® Gel for the Reduction of Scar Formation in Surgical Wounds Following Bilateral Anchor Incision Breast Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xequel Bio, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-SCAR-01
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Mammoplasty; Scarring; Scar; Breast Reconstruction
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Granexin® gel 100 μM (Experimental): Within-subject comparison of Granexin® Gel versus vehicle gel (placebo).
  Granexin® gel 100 μM will be applied four times over three days: twice during surgery, 24 hours after surgery and 48 hours after surgery. Granexin® will be applied on the right or left breast according to a randomization list.
  Interventions: Drug: Granexin® gel 100 μM; Drug: Vehicle gel
- Granexin® gel 200 μM (Experimental): Within-subject comparison of Granexin® Gel versus vehicle gel (placebo).
  Granexin® gel 200 μM will be applied four times over three days: twice during surgery, 24 hours after surgery and 48 hours after surgery. Granexin® will be applied on the right or left breast according to a randomization list.
  Interventions: Drug: Granexin® gel 200 μM; Drug: Vehicle gel
- Vehicle Gel (Placebo Comparator): Within-subject comparison of Granexin® Gel versus vehicle gel (placebo).
  Vehicle gel will be applied four times over three days: twice during surgery, 24 hours after surgery and 48 hours after surgery. Granexin® will be applied on the right or left breast according to a randomization list.
  Interventions: Drug: Granexin® gel 100 μM; Drug: Granexin® gel 200 μM; Drug: Vehicle gel

INTERVENTIONS:
Drug: Granexin® gel 100 μM — Administered during the surgery, 24 hours post-surgery, and 48 hours post-surgery.
  Arms: Granexin® gel 100 μM; Vehicle Gel
Drug: Granexin® gel 200 μM — Administered during the surgery, 24 hours post-surgery, and 48 hours post-surgery.
  Arms: Granexin® gel 200 μM; Vehicle Gel
Drug: Vehicle gel — Administered during the surgery, 24 hours post-surgery, and 48 hours post-surgery.
  Other Names: placebo

SUMMARY:
The purpose of this study is to evaluate effectiveness of Granexin® gel in reducing scar formation in surgical incisional wounds.

DETAILED DESCRIPTION:
Participants that meet screening criteria will be eligible for randomization providing all other criteria are met. Participants enrolled will receive study drug for 3 days. The participants will have an additional follow-up period to assess scarring of both Granexin® gel and Vehicle gel incisions through end of study at Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 18 years and older
2. Female subjects of childbearing potential must have a negative urine or blood pregnancy test at screening and baseline.
3. Female subjects of childbearing potential must agree to use ONE of the following birth control methods throughout the study:

   * abstinence
   * condom with spermicide
   * diaphragm with spermicide
   * Hormonal contraceptive
   * intra-uterine device

   Non-childbearing confirmed by prior documentation of at least one of the following:
   * postmenopausal
   * surgically sterilized
4. Subjects undergoing a breast surgery procedure with bilateral anchor incisions
5. Signed informed consent form

Exclusion Criteria:

1. Subjects with breast implants or history of breast implants
2. Subjects undergoing breast surgery requiring breast implants
3. Subjects requiring nipple grafting using any technique
4. Subjects with a history of infection in the past 6 months in the intended area of incision
5. Subjects with breast tattoos in the intended area of the incision
6. Subjects with known skin sensitivity to Tegaderm™
7. Subjects with a history of keloids
8. Known conditions of collagen vascular diseases
9. Subjects with clinically significant medical conditions as determined by the Investigator, which would impair wound healing including renal, hepatic, hematologic, neurologic or autoimmune disease. Examples include but are not limited to:

   1. Renal insufficiency as an estimated GFR, which is < 30 mL/min/1.7m2
   2. Abnormal blood biochemistry defined as 3 times that of the upper limit of the normal range
   3. Hepatic insufficiency defined as total bilirubin > 2 mg/dL or serum albumin < 25 g/L
   4. Hemoglobin < 9 g/dL
   5. Hematocrit < 30%
   6. Platelet count < 100,000 μL
10. Any history within the last 5 years or the presence of any active systemic cancer (with the exception of non-melanoma skin cancer)
11. Current treatment with systemic corticosteroids (>15 mg/day). Washout period is 30 days prior to screening
12. Current treatment with biologic immunosuppressive agents or chemotherapeutic agents. Wash out period for short term immunosuppressive agents is 14 days prior to screening
13. Previous history of radiation therapy to the chest
14. Known inability to complete required study visits during study participation
15. A psychiatric condition (e.g., suicidal ideation), chronic alcohol consumption, or drug abuse problem determined from the subject's medical history, which, in the opinion of the Investigator, may pose a threat to subject compliance
16. Use of any investigational drug or therapy within the 28 days prior to screening
17. History of previous breast surgeries in the area where the incisions are to be made
18. Currently pregnant, pregnant during the 6 months prior to screening, lactating, or breastfeeding
19. Any other factor, which may, in the opinion of the Investigator, compromise participation and follow-up in the study
20. Any areolar abnormalities that are deemed clinically significant by the Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Change in scar severity at Month 12 | Month 12
  Assessed using the Patient and Observer Scar Assessment Scale (POSAS). The POSAS has a rage from 6 to 60 with higher scores indicating worse outcomes. One scale will be used for each segment of the scar. The score from each segment will be combined into one score.

SECONDARY OUTCOMES:
Change in scar severity at Month 6, Month 9 and Month 12 | Month 6, Month 9 and Month 12
  Assessed using the Scar Cosmesis Assessment and Rating (SCAR) Scale. The SCAR scale has a range of 0 (best possible scar) to 15 (worst possible scar).
Change in scar severity at Month 9 | Month 9
  Assessed using the Patient and Observer Scar Assessment Scale (POSAS). The POSAS has a range from 6 to 60 with higher scores indicating worse outcomes. One scale will be used for each segment of the scar. The score from each segment will be combined into one score.
Proportion of subjects with incision healing complications | Day 1 to Month 12
  Investigator's assessment of incision healing complications
Proportion of subjects with incision infection | Day 1 to Month 12
  Investigator's assessment of presence or absence of infection

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Private Clinic- David Kulber, Los Angeles, California
  - Pasadena Surgeons, Pasadena, California
  - Universal Axon Clinical Research, Doral, Florida
  - Miami Plastic Surgery, Miami, Florida
  - Ibrahim H. Amjad, MD, PA, West Miami, Florida
  - Northwestern University - Feinberg School of Medicine - Division of Plastic & Reconstructive Surgery, Chicago, Illinois
  - Iowa Plastic Surgery, Davenport, Iowa
  - Luxurgery, New York, New York
  - Wake Forest Baptist Hospital - Plastic and Reconstructive Surgery, Winston-Salem, North Carolina
  - Integrated Aesthetics, Spring, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No